CLINICAL TRIAL: NCT00210925
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Flexible Dose Study to Assess the Safety and Efficacy of Topiramate in the Treatment of Alcohol Dependence
Brief Title: An Efficacy and Safety Study of Topiramate in the Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004681
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Alcoholism
Keywords: alcoholism; alcohol dependence; medication treatment.
MeSH Terms: conditions — Alcoholism | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of topiramate compared to placebo in patients with alcohol dependence.

DETAILED DESCRIPTION:
The impact of alcoholism can be reduced through effective treatments, which may include medical, psychological, and social interventions. The main goals of alcohol-dependence treatment are to assist patients in avoiding alcohol, developing better strategies for managing stress, and improving self-esteem and quality of life. Studies have demonstrated that treatments for alcohol use disorders can be effective, but their effectiveness is often limited. Although the optimal goal of treatment should be total abstinence, even patients who are unable to achieve this goal may still benefit from treatments leading to a reduction in drinking. Medications are commonly used in other addictive disorders, such as nicotine and opioid dependence, suggesting that this intervention could be useful in the treatment of alcohol dependence. This is a randomized, double-blind, flexible dose study to determine if topiramate, a prescription medication approved by the Food & Drug Administration for the treatment of epilepsy and the prevention of migraine, administered at a dose of 300mg per day or the subject's maximum tolerated dose, is safe and effective compared with placebo in patients with alcohol dependence. The study hypothesis is that topiramate will be more effective than placebo in reducing the percentage of heavy drinking days (5 or more standard drinks per day for men and 4 or more standard drinks per day for women) in patients with alcohol dependence. The patients will receive topiramate tablets (25mg and/or 100mg) or matching placebo. Study medication is taken in increasing doses starting at 25 mg/day up to 300 mg per day (or maximum tolerated dose) during the first 6 weeks and the achieved dose is maintained for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of alcohol dependence
* drink an average of 28 or more standard drinking units/week for women or 35 or more standard drinking units/week for men
* have a desire to stop drinking completely or to reduce alcohol consumption with the possible long-term goal of abstinence
* have a body mass index of 18 or more
* sexually active women capable of having children must be using an acceptable method of birth control
* must be in generally good health.

Exclusion Criteria:

* No current or recent (within 6 months) diagnosis of other substance abuse or dependence
* no inpatient or outpatient counseling for alcohol dependence other than Alcoholics Anonymous within 4 weeks
* not more than 4 past failed inpatient treatments attempts for alcohol dependence
* no other psychiatric disorder that requires treatment with medication or therapy
* no current probation or parole requirement or legally mandated requirement to participate in an alcohol treatment program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2004-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The change in percentage of heavy drinking days (5 or more standard drinking units per day for men and 4 or more standard drinking units per day for women) from baseline at 12 weeks or final visit.

SECONDARY OUTCOMES:
The change in each of the following: drinks/drinking day, drinks/day, percent days abstinent, Clinical Institute Withdrawal Assessment for Alcohol-revised, compared to baseline at 12 weeks or final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Johnson BA, Rosenthal N, Capece JA, Wiegand F, Mao L, Beyers K, McKay A, Ait-Daoud N, Anton RF, Ciraulo DA, Kranzler HR, Mann K, O'Malley SS, Swift RM; Topiramate for Alcoholism Advisory Board; Topiramate for Alcoholism Study Group. Topiramate for treating alcohol dependence: a randomized controlled trial. JAMA. 2007 Oct 10;298(14):1641-51. doi: 10.1001/jama.298.14.1641. PMID 17925516
- [Derived] Falk DE, O'Malley SS, Witkiewitz K, Anton RF, Litten RZ, Slater M, Kranzler HR, Mann KF, Hasin DS, Johnson B, Meulien D, Ryan M, Fertig J; Alcohol Clinical Trials Initiative (ACTIVE) Workgroup. Evaluation of Drinking Risk Levels as Outcomes in Alcohol Pharmacotherapy Trials: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Psychiatry. 2019 Apr 1;76(4):374-381. doi: 10.1001/jamapsychiatry.2018.3079. PMID 30865232
- [Derived] Johnson BA, Rosenthal N, Capece JA, Wiegand F, Mao L, Beyers K, McKay A, Ait-Daoud N, Addolorato G, Anton RF, Ciraulo DA, Kranzler HR, Mann K, O'Malley SS, Swift RM; Topiramate for Alcoholism Advisory Board; Topiramate for Alcoholism Study Group. Improvement of physical health and quality of life of alcohol-dependent individuals with topiramate treatment: US multisite randomized controlled trial. Arch Intern Med. 2008 Jun 9;168(11):1188-99. doi: 10.1001/archinte.168.11.1188. PMID 18541827
- See also: Topiramate vs. Placebo in Alcohol Dependence — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=621&filename=CR004681_CSR.pdf